CLINICAL TRIAL: NCT02830516
Title: Intraoperative Measurement of Lung Elastance and Transpulmonary Pressure Using Two Different Methods
Acronym: Lungbaro
Status: Completed | Type: Observational
Sponsor: Stefan Lundin (Other)
Responsible Party: Sponsor-Investigator, Stefan Lundin, Professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: LUA-74201
Record Dates: First submitted 2016-06-21; First posted 2016-07-13 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung elastance - transpulmonary pressure: Lung elastance and transpulmonary pressure measured by tidal esophageal pressure variations and by performing a PEEP step
  Interventions: Other: Measurement of lung elastance by two methods

INTERVENTIONS:
Other: Measurement of lung elastance by two methods — Measurement of tidal variations in esophageal pressure followed in the same patient by performing a PEEP-step while simultaneously measuring the change in lung volume

SUMMARY:
Classically lung elastance and transpulmonary pressure are measured from the difference in tidal variations of airway pressure subtracted by tidal variations i esophagus pressure divided by the tidal volume. This requires the presence of a esophageal balloon catheter which is cumbersome and costly. In this study values obtained as described above are compared to values obtained with a new method in which a stepwise increase in positive endexpiratory pressure (PEEP) is performed with a size which corresponds to the tidal volume which the patient is ventilated with. These measurements are performed in anesthetized patients prior to major surgery.

DETAILED DESCRIPTION:
Classically lung elastance and transpulmonary pressure are measured from the difference in tidal variations of airway pressure subtracted by tidal variations in esophageal pressure divided by the tidal volume (Method 1). This requires the presence of a esophageal balloon catheter which is cumbersome and costly.

In this study values obtained as described in Method 1 above are compared to values obtained with a new method in which a PEEP-step is performed with a size which corresponds to the tidal volume which the patient is ventilated with. Measurements using Method 1 and 2 are performed in anesthetized patients prior to major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major surgery during anesthesia and muscle relaxation

Exclusion Criteria:

* Patient with chronic obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients which are anesthetized and muscle relaxed and are planned to undergo major surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of lung elastance | At 1 hour
  Comparison of two method for measurements of lung elastance (Measurement of tidal variations in esophageal pressure followed in the same patient by performing a PEEP-step while simultaneously measuring the change in lung volume)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, Professor, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Persson P, Stenqvist O, Lundin S. Evaluation of lung and chest wall mechanics during anaesthesia using the PEEP-step method. Br J Anaesth. 2018 Apr;120(4):860-867. doi: 10.1016/j.bja.2017.11.076. Epub 2017 Dec 1. PMID 29576127